CLINICAL TRIAL: NCT02460796
Title: Hippotherapy on Functional Capacity and Quality of Life in Parkinson's Disease: a Prospective Study
Brief Title: Hippotherapy and Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: University of Brasilia (Other)
Collaborators: Wilfrid Laurier University (Other)
Responsible Party: Principal Investigator, Rita de Cassia Pereira Pinto Homem MSc, MSc, University of Brasilia
Other Study IDs: UnBrasilia
Record Dates: First submitted 2015-05-26; First posted 2015-06-02 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Quality of Life; Parkinson's Disease
Keywords: Parkinson's disease; Quality of life; Gait velocity; Capacity
MeSH Terms: conditions — Parkinson Disease | interventions — Equine-Assisted Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Weeks
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- hippotherapy group or study group: 8 weeks of hippotherapy therapy: Familiarization sessions were initially 15 minutes and gradually evolved to 30 minutes in order to allow all participants to adapt to the horse's rhythmic movements and to the act of mounting the horse. Each session had warm up before the training and exercises for relaxation in the end of each session.
  Interventions: Other: Hippotherapy
- control group: 8 weeks of Parkinson's disease lectures: this group did not hippotherapy classes in the same period.

INTERVENTIONS:
Other: Hippotherapy — The sessions began with a 5 minutes warm up that involved stretching and body awareness exercises. Then, the training was conducted for 20 minutes with arms and torso exercises, changes of direction called serpentine movements; up and down hip movements with feet on stirrups, and forced expiration. In the final 5 minutes, exercises for relaxation were conducted with the horse which involved moving the hand on the horse's neck, laying forward on the head and stroking the horse. The horses walking speed was between 5.8 and 6.4 Km/h.
  Other Names: Equine Therapy
  Groups: hippotherapy group or study group

SUMMARY:
BACKGROUND: Motor symptoms associated with Parkinson's disease may impair one's independence and ability to perform daily activities consequently decreases quality of life. Hippotherapy has been shown as an effective treatment to improve function in daily activities and quality of life in other neurological populations, thus a study was conducted to assess the effects of hippotherapy in people with Parkinson's disease.

METHODS: Nine volunteers formed the treatment group which participated in a ten-week hippotherapy program, and nine individuals formed the control group (attended a ten-week series of lessons on Parkinson's disease). Outcome measures included 30-second chair stand (as a measure of strength-endurance), gait velocity (during 10m walk test) and health-related quality of life.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is associated with motor symptoms such as bradykinesia, rigidity and postural instability 1 which interfere with the patient's independence, and ability to carry out activities of daily life 2. In addition, losses in functional may result in a decreased health-related quality of life (HRQL) 3. Thus, as PD progresses HRQL gets worse 4.

Exercise programs are suggested to improve functional capacity and HRQL in people with PD 3. However, in the later stages of PD, mobility problems restrict the potential to participate in exercise programs, resulting in even greater loss in functional capacity and HRQL. Furthermore, a decline in the efficacy of pharmacological treatment and complications due to motor fluctuations and medication side effects make the role of complementary treatments such as hippotherapy critical to individuals with PD at late stages. Hippotherapy is a therapeutic intervention commonly used in populations with mobility deficits, since they do not require effort or walking from patients who can no exercise in standing position. When is on the horse, the patient exercises as he/she is walking unassisted 5. Neurological conditions are improved by horse's movement stimulations. The set formed by the patient and his horse performs rhythmic and three-dimensional oscillations which trigger very important neuromuscular responses from the rider's postural reflex mechanisms 6. The horse's movements are sensed by the participant on the saddle, and when the horse is slowly walking it has been argued to be similar to the pelvic movement produced by human gait, thereby strengthening the trunk muscles and improving balance 7. The senses are integrated during the act of riding performing sensory stimulation 8. Furthermore, hippotherapy has been demonstrated to be an effective method to improve functional capacity by increasing gait velocity in people with brain disorders 9, functional mobility in elderly 10 and functional strength in people after stroke 11 and in people with spinal cord injury 5. In addition, hippotherapy has been shown to improve HRQL in children and in adults 6.

Considering the potential benefits of hippotherapy to anticipatory postural adjustments and sensory stimulation 9, 11, it could be hypothesized that hippotherapy may increase functional capacity and improve HRQL in individuals with PD. This hypothesis has not been tested yet. Therefore, the purpose of this study was to assess the effects of a hippotherapy program on functional capacity and on HRQL in people with PD.

(4) Methods

Subjects People with confirmed diagnosis of PD by medical report were invited through advertisements on radio, on television, public announcements and posters around the hospitals to participate in the Physical Activities Program for Persons with Neurodegenerative Diseases. Among 81 registered volunteers, 18 participants, six women and twelve men, unable to perform usual physical activity because they were in the late stages according to Hoehn and Yahr scale (H & Y≥ 3), or because they need to use a wheelchair for severe mobility problems were enrolled in the hippotherapy program which formed the sample (n=18). Exclusion criteria were uncontrolled hypertension, unstable cardiovascular disease and had practiced riding or hippotherapy six months before the intervention period. Among the 18 volunteers from the sample, three women and six men were randomized for the intervention group called hippotherapy group (HT) (n=9), which performed ten weeks of hippotherapy sessions (2 familiarization + 8 hippotherapy weeks) twice a week with each session lasting thirty minutes. Nine other participants who were waiting to be allocated to the hippotherapy program in the following semester attended lectures on PD, twice a week for ten weeks, with each session lasting thirty minutes. Demographics and characteristics of the sample can be seen in Table 1. This study was approved by the Research Ethics Committee of the University of Brasilia on 10/10/2013 by the number CAAE 17329213.7.0000.0030. All participants were informed about the procedures and agreed to participate in the study signing the informed consent term.

Instruments Quality of life was measured using the Parkinson's Disease Quality of Life Questionnaire (PDQL) Brazilian version 4.

Functional mobility was evaluated by the Timed Up and Go Test (TUG) according Podsiadlo and Richardson 12.

Strength endurance was measured using the Thirty-second Chair Stand Test (30CST) according Gill and McBurney 13.

Gait velocity was evaluated using the Ten Meter Walk Test (TMW) according Bohannon, Andrews and Thomas 14.

All functional tests had three trials with a 2 minutes interval between each trial, and the average of the two last measurements was used for analysis.

Hippotherapy Procedures Familiarization sessions were initially 15 minutes and gradually evolved to 30 minutes in order to allow all participants to adapt to the horse's rhythmic movements and to the act of mounting the horse. The sessions were performed at the First Regiment of Cavalry Guard of the Brazilian Army. All practitioners used helmet, shirt, pants and closed shoes. The team was composed by an auxiliary guide, a physical education teacher and two auxiliaries. In order to mount and dismount, all participants used a specific ramp for hippotherapy classes. All horses used saddle and riding equipment, the stirrups were individually adjusted.

The sessions began with a 5 minutes warm up that involved stretching and body awareness exercises. Then, the training was conducted for 20 minutes with arms and torso exercises, changes of direction called serpentine movements; up and down hip movements with feet on stirrups, and forced expiration. In the final 5 minutes, exercises for relaxation were conducted with the horse which involved moving the hand on the horse's neck, laying forward on the head and stroking the horse. The horses walking speed was between 5.8 and 6.4 Km/h.

In order to assess the effect of the hippotherapy the difference between post and pre-tests scores for each dependent measure was calculated (delta (∆)).

To assess whether data had normal distribution the Shapiro-Wilk test was used, which did not indicate a normal distribution for functional capacity variables. Thus, the Mann-Whitney U test for independent samples was used in order to compare the changes in functional capacity between groups. The Shapiro-Wilk test demonstrated a normal distribution for PDQL variables data, and then parametric statistics was performed with a one-way analysis of variance (ANOVA). Statistical analysis was performed using the program Statistica 7.0 (StatSoft Inc., Tulsa, Oklahoma, USA), adopting a significance level of p≤0.05.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease patient with H&Y level 3 at least

Exclusion Criteria:

* Uncontrolled hypertension, unstable cardiovascular disease, chronical disease that can invalidate the research and had practiced riding or hippotherapy six months before the intervention period.

Ages: 65 Years to 83 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: 18 volunteers with Parkinson's desease.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2013-06; Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Increment of gait speed | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rita C Homem, MSc, Principal Investigator — UnB; Ricardo J Oliveira, PhD, Study Director — UnB

REFERENCES:
- [Background] Han JY, Kim JM, Kim SK, Chung JS, Lee HC, Lim JK, Lee J, Park KY. Therapeutic effects of mechanical horseback riding on gait and balance ability in stroke patients. Ann Rehabil Med. 2012 Dec;36(6):762-9. doi: 10.5535/arm.2012.36.6.762. Epub 2012 Dec 28. PMID 23342307
- [Background] Lee CW, Kim SG, Yong MS. Effects of hippotherapy on recovery of gait and balance ability in patients with stroke. J Phys Ther Sci. 2014 Feb;26(2):309-11. doi: 10.1589/jpts.26.309. Epub 2014 Feb 28. PMID 24648655
- [Background] de Araujo TB, de Oliveira RJ, Martins WR, de Moura Pereira M, Copetti F, Safons MP. Effects of hippotherapy on mobility, strength and balance in elderly. Arch Gerontol Geriatr. 2013 May-Jun;56(3):478-81. doi: 10.1016/j.archger.2012.12.007. Epub 2013 Jan 3. PMID 23290005
- [Background] Janura M, Peham C, Dvorakova T, Elfmark M. An assessment of the pressure distribution exerted by a rider on the back of a horse during hippotherapy. Hum Mov Sci. 2009 Jun;28(3):387-93. doi: 10.1016/j.humov.2009.04.001. Epub 2009 Apr 29. PMID 19406498
- [Background] Lechner HE, Kakebeeke TH, Hegemann D, Baumberger M. The effect of hippotherapy on spasticity and on mental well-being of persons with spinal cord injury. Arch Phys Med Rehabil. 2007 Oct;88(10):1241-8. doi: 10.1016/j.apmr.2007.07.015. PMID 17908564